CLINICAL TRIAL: NCT02904122
Title: Validation Study of Oral Teleconsultation
Brief Title: Oral Teleconsultation
Acronym: EDENT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9173
Record Dates: First submitted 2016-09-07; First posted 2016-09-16 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2013-06

CONDITIONS: Dental Care
MeSH Terms: interventions — Remote Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Teleconsultation (Other): Teleconsultation using a specific camera SoproCare®6
  Interventions: Other: teleconsultation

INTERVENTIONS:
Other: teleconsultation — Determine the interest of teleconsultation in dentistry tool for the diagnosis of caries. Ie whether oral teleconsultations are of the same quality as conventional consultations for the diagnosis of caries ..

SUMMARY:
In this study we want to compare a dental diagnose during face to face consultation vs remote consultation with telemedicine device.

DETAILED DESCRIPTION:
Using Soprocare® camera, videos of patients' oral cavity are recorded and analysed remotely. 200 patients have been included: 100 in Montpellier (France) and 100 in Kitakyushu (Japan).

A classical face-to-face oral consultation is realized using ICDAS II classification. Then a student recorded 6 videos of patients' mouth: one video by sector, showing each face of molars and premolars in cario fluorescence mode of Soprocare® and one video of the maxillary and mandibular incisor-canine block in perio mode.

In a third step, a remote dentist analysed videos and made a telediagnosis using the same classification. Dental hygiene and missing teeth are also noted in classical and tele diagnostic.

The direct and the tele diagnostic are compared.

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged at least 18 years
* The subject must be given free and informed consent
* Topics scheduled consultation from the dental center of Montpellier University Hospital and the Center Kyushu University (Japan).

Exclusion Criteria:

* NA

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
diagnostic of caries | 1 day
  Teleconsultation will be made using a specific camera SoproCare®6, the company Acteon ..

IPD SHARING:
Plan to Share IPD: Undecided